CLINICAL TRIAL: NCT06680973
Title: Comparison of the Effects of Hospital-Based and Home-Based Resistance Training in Individuals with Adult Congenital Heart Disease
Brief Title: Hospital-Based and Home-Based Resistance Training in Adult Congenital Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Topcuoglu, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/09-11
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Diseases; Resistance Training; Muscle Strength; Functional Capacity
Keywords: Congenital Heart Diseases; Resistance training; Muscle strength; Functional capacity
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial design will be employed. Block randomization will be performed using computer-assisted randomization software (https://www.graphpad.com/quickcalcs/randomize1/), and stratified randomization will be applied to ensure equal gender distribution across groups. Participants will be divided into three groups:
  Hospital-based resistance training group Home-based resistance training group Control group
  The individuals in the hospital-based and home-based resistance training groups will undergo a 12-week training program, with evaluations conducted twice: once before and once after the training. In the control group, no training will be provided, and evaluations will be performed twice, with a 12-week interval between assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hospital-Based Resistance Training Group (Experimental): Participants will undergo resistance training using a weight training station and elastic equipment (elastic bands and tubes).
  Interventions: Other: Hospital-Based Resistance Training
- Home-Based Resistance Training Group (Experimental): Participants will undergo resistance training at home using elastic equipment (elastic bands and tubes).
  Interventions: Other: Home-Based Resistance Training
- Control Group (No Intervention): No training will be provided to the participants.

INTERVENTIONS:
Other: Hospital-Based Resistance Training — Participants will undergo resistance training using a weight training station and elastic equipment (elastic bands and tubes).
  The intensity of the resistance training with the weight training station will be determined based on 1 Repetition Maximum (1RM). Resistance training with the weight training station will be conducted at 30-70% of the 1RM intensity and will include the following exercises: leg extension, pull down, chest press, and pec deck.
  The intensity of resistance training using elastic equipment will be determined according to the individual's perceived exertion. Resistance training with elastic equipment will be performed at an intensity of 12-14 on the Borg Scale (moderate to somewhat hard) for movements involving hip flexion, extension, abduction, and adduction.
  The resistance training regimen will consist of 8-12 repetitions, 2-3 sets, with at least 1 minute of rest between sets, twice a week for 12 weeks.
  Arms: Hospital-Based Resistance Training Group
Other: Home-Based Resistance Training — Participants will undergo resistance training at home using elastic equipment (elastic bands and tubes). The intensity of the resistance training will be determined based on the individual's perceived exertion. The training will be conducted at an intensity of 12-14 on the Borg Scale (moderate to somewhat hard), with 8-12 repetitions, 2-3 sets, and a rest period of at least 1 minute between sets, twice a week for 12 weeks. Progression in training intensity will be achieved by increasing the weight once the perceived exertion, as measured on the Modified Borg Scale, falls below 3 (moderate) after completing 20 repetitions.
  Resistance training will include exercises such as leg extension, pull down, chest press, pec deck, and movements involving hip flexion, extension, abduction, and adduction. To ensure individuals perform exercises correctly, follow-up will be conducted through online meetings every two weeks. These meetings will not be recorded.
  Arms: Home-Based Resistance Training Group

SUMMARY:
Congenital heart disease (CHD) is defined as functional or anatomical abnormalities of the heart and major intrathoracic vessels present at birth. Impaired responses to exercise in individuals with CHD reduce exercise capacity and increase long-term mortality risk. Today, the growing population of adults with congenital heart disease (ACHD) faces chronic issues stemming from congenital abnormalities, along with muscle strength loss and a decline in activities of daily living. Once the planned treatments in this project proposal are implemented and data are obtained (especially if these data support the hypotheses), the treatment protocols applied in this study and their effects will be considered alongside the current treatment plans for individuals with CHD who experience muscle strength loss and disease-related impairment. With new treatment programs, this study aims to reduce disease-related muscle strength loss, improve disease-related outcomes, and enhance quality of life.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is defined as congenital functional or anatomical abnormalities of the heart and the major intrathoracic vessels. There are numerous physiological changes that accompany and facilitate the circulatory system's adaptation to the hemodynamic demands of exercise. In individuals with CHD, altered cardiovascular anatomy and physiology adversely affect responses to exercise in various ways and to varying degrees. Impairment in in individuals with CHD reduces exercise capacity and increases long-term mortality risk. The impairment in responses to exercise makes the prescription and progression of exercise challenging. Nowadays, the increasing lifespan of the adult congenital heart disease (ACHD) population faces not only chronic issues stemming from congenital abnormalities but also muscle strength loss and a reduction in daily living activities. Early assessment of muscle strength and exercise capacity in individuals with ACHD and the implementation of appropriate exercise training will reduce the incidence of all cause and cardiovascular disease mortality. Despite the increased disease related impact and mortality risk associated with age in individuals with CHD, the number of studies on individuals with ACHD is insufficient compared to studies conducted on children.

It has been shown that resistance exercise, similar to aerobic exercise, improves symptomatic responses and responses to exercise; and can be safely applied in individuals with CHD. In cardiovascular diseases, resistance training not only maintains and increases muscle strength and mass but also has positive physiological and clinical effects on the cardiovascular system and risk factors. There are also studies showing that resistance training improves daily living activities and quality of life. The use of different application models in cardiac rehabilitation is becoming increasingly widespread. Today, increased healthcare expenditures and economic problems have emphasized the importance of minimal equipment requirements. Minimal equipment requirements, a widely accessible patient group, and reduced transportation issues and costs highlight the importance of home-based cardiac rehabilitation.

The study is designed to be prospective, randomized, and double-blind. Participants will be divided into three groups: a hospital-based resistance training group, a home-based resistance training group, and a control group. At least 33 individuals with CHD (at least 11 individuals per group) will be included in the study. The long-term effects of the exercise will be assessed using the following: peripheral muscle strength with a manual muscle testing device, functional capacity with the six-minute walk test, daily living activities with the Glittre Daily Living Activities Test, upper extremity exercise capacity with the six minute Pegboard and Ring Test, arterial stiffness with an oscillometer-based device using the pulse wave velocity technique. Participants will undergo hospital-based resistance training in one group and home-based resistance training in the other group, twice a week for 12 weeks. No training will be provided to the control group. Assessments will be conducted twice, before and after the exercise training.

Once the planned treatments in the project proposal are implemented and data is obtained, the treatment protocols and their effects applied within the scope of the study will also be considered for individuals with CHD included in the study and for those diagnosed with CHD who experience disease-related exposure and muscle strength loss after the project. The new treatment programs aim to reduce disease-related exposure and muscle strength loss and to improve quality of life. It is planned to prepare research articles and international conference presentations from the data obtained from the project.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital heart disease
* Aged between 18 and 45 years
* Being informed about the study and providing written consent to participate
* Clinical stability has been achieved in the patients
* No changes in ongoing medication treatment that negatively affect clinical stability

Exclusion Criteria:

* Having additional cardiovascular, neurological, orthopedic, or any other systemic diseases
* Being classified as high risk (severe systolic dysfunction, moderate/severe elevated pulmonary artery pressure, significant arrhythmic burden, malignant arrhythmia, etc.)
* Not suitable for cognitive, psychological, and mental assessments
* Undergoing a surgery other than heart surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
Peripheral Muscle Strength- Isotonic | From immediately before the treatment began to 12 weeks after the treatment.
  Isotonic strength will be assessed three times on both the right and left sides. Isotonic strength will be evaluated using the 1-repetition maximum technique with a weight training station for knee extension, pull down, chest press, and pec deck functions.
Peripheral Muscle Strength-Isometric | From immediately before the treatment began to 12 weeks after the treatment
  Isometric strength will be assessed three times on both the right and left sides. Isometric strength will be assessed using a manual muscle testing device (K-Force Push, France) for knee extension, shoulder and hip abduction, flexion, and extension, as well as elbow flexion and extension.
Hand Grip Strength | From immediately before the treatment began to 12 weeks after the treatment.
  Maximum isometric hand grip strength will be assessed using a digital hand dynamometer (K-Force Grip, France). During the test, individuals will be seated upright in a chair with their elbow positioned at a 90° flexion. Three measurements will be taken for both the right and left hands, and the highest value will be recorded. A 20-second rest period will be allowed between measurements.
Functional Capacity | From immediately before the treatment began to 12 weeks after the treatment.
  Functional capacity will be assessed using the 6-minute walk test (6 MWT). For the 6 MWT, the start and end points of a 30-meter corridor will be marked, and participants will be instructed to walk the distance at their maximum walking speed without running for 6 minutes. Before and after the test, fatigue levels will be recorded using the Borg scale, along with measurements of blood pressure, heart rate, and oxygen saturation. The 6 MWT is considered an easily applicable, widely used, and safe submaximal exercise test for individuals with congenital heart disease.
Activities of Daily Living (ADL) | From immediately before the treatment began to 12 weeks after the treatment.
  The Glittre Activities of Daily Living (ADL) Test will be used to assess activities of daily living and functional status. Participants will begin the test in a seated position, wearing backpacks weighing 5 kg for men and 2.5 kg for women. The test will take place over a 10-meter distance between a chair and a shelf, with a two-step staircase located in the middle. Participants will be asked to walk as quickly as possible to the steps, climb up and down, pick up a 1-kilogram bottle from the shelf, first place it in the center, then lower it, return it to the center, and finally place it at the top. They will then return, pass the steps, sit back in the chair, and stand up again to complete one round. The total time taken to complete five rounds will be recorded in minutes.
Upper Extremity Exercise Capacity | From immediately before the treatment began to 12 weeks after the treatment.
  The Six-Minute Pegboard and Ring Test (6-PBRT) will be used to assess upper extremity exercise capacity. For the test, a board will be used with six holes spaced 10 cm apart on a horizontal plane, and six additional holes will be positioned 20 cm below them in alignment. Four wooden rods, easily inserted and removed from the holes, will be placed, and 20 rings that fit the rods will be used. The placement of the rods will be based on the individual's shoulder width measurement. Participants will be instructed to place the rings with both hands, first from the bottom to the top, then from the top to the bottom, over the course of six minutes. Two rings that are removed and replaced simultaneously will be counted as one set. At the end of the six minutes, the total number of rings placed will be recorded in terms of the number of completed rings.
Body Composition | From immediately before the treatment began to 12 weeks after the treatment.
  The lean body mass percentage of the individual will be determined by Bioelectrical Impedance Analysis. The measurement will be made by the individual standing on the device with bare feet and waiting. If the lean body mass percentage values are in the normal range, the body composition is normal; lean body mass percentage low values indicate deterioration of body composition.
Arterial Stiffness | From immediately before the treatment began to 12 weeks after the treatment.
  Arterial stiffness will be assessed non-invasively using the Mobil-O-GRAPH (TG) device (I.E.M., Stolberg, Germany), an oscillometer-based device, with the pulse wave velocity (PWV) technique. During the measurement, the patient will sit in an upright position on a chair and remain still in silence. The cuff of the device will be placed on the individual's right arm, with its lower edge positioned above the elbow. The individual's arm will be supported and fixed with a pillow to align with the level of the heart.

SECONDARY OUTCOMES:
Functional Mobility | From immediately before the treatment began to 12 weeks after the treatment.
  It will be evaluated using the 4-meter Walk Test. The 4-meter walk test will be conducted on a 4-meter long track, with clearly marked start and end points using cones. The patient will be asked to complete the test at their usual walking speed. The timer will start at the initial movement and stop when the end point is crossed.
Functional Mobility with Dual Task | From immediately before the treatment began to 12 weeks after the treatment.
  It will be evaluated using the Dual-Task Timed Up and Go Test.The Dual-Task Timed Up and Go Test, individuals will be asked to stand up from a chair, walk 3 meters at a safe and normal pace, turn around, walk back, and sit down again, with the time recorded in seconds. During the test, individuals will also be asked to hold a glass of water in one hand to assess motor function, and to count backward from 100 in threes to assess cognitive function. A shorter time indicates better balance and mobility ability.
Cognition | From immediately before the treatment began to 12 weeks after the treatment.
  It will be evaluated using the Montreal Cognitive Assessment (MoCA) test. The MoCA assesses functions such as short-term memory, visuospatial skills, executive functions, abstract thinking, verbal fluency, attention, concentration, and language. The highest possible total score on the test is 30. The normal cut off score for the test is 21 points or higher. The Turkish validity and reliability of the scale were conducted by Ozdilek et al.
Health-Related Quality of Life | From immediately before the treatment began to 12 weeks after the treatment.
  It will be assessed using the Short Form-36 (SF-36). The SF-36 is a scale that evaluates general health perception and quality of life. It consists of a total of 8 subcategories: physical function, role limitations due to physical problems, role limitations due to emotional problems, vitality, social functioning, pain, and general health perception. The scale includes 36 items and 11 questions. Each subcategory is scored between 0 and 100. A higher score indicates a higher quality of life. The Turkish validity and reliability of the scale were conducted by Pinar et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niedermeyer CDC, Shizukuishi MLY, Schaan CW, Lukrafka JL. Peripheral and respiratory muscle strength in children and adolescents with CHD: systematic review and meta-analysis. Cardiol Young. 2022 Nov;32(11):1728-1741. doi: 10.1017/S1047951122003092. Epub 2022 Oct 6. PMID 36200343
- [Background] Bernier PL, Stefanescu A, Samoukovic G, Tchervenkov CI. The challenge of congenital heart disease worldwide: epidemiologic and demographic facts. Semin Thorac Cardiovasc Surg Pediatr Card Surg Annu. 2010;13(1):26-34. doi: 10.1053/j.pcsu.2010.02.005. PMID 20307858